CLINICAL TRIAL: NCT05989750
Title: Air-polishing With Erythritol on Prevalence of White Spot Lesions and Gingivitis During Orthodontic Treatment With Fixed Appliances: a Randomized Clinical Trial of 2-years Duration
Brief Title: Air-polishing With Erythritol During Orthodontic Tretament
Acronym: AirPort
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Catherine Giannopoulou (Other)
Collaborators: University of Geneva, Switzerland (Other)
Responsible Party: Sponsor-Investigator, Catherine Giannopoulou, Professor, University of Geneva, Switzerland
Organization: University of Geneva, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BASEC 2023-D0032
Record Dates: First submitted 2023-07-14; First posted 2023-08-14 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Inflammation Gum; White Spot Lesion
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Intervention Model Description: Randomized, examiner-masked clinical trial
Who Masked: Investigator
Masking Description: The examiner, the biostatistician and people working in the laboratory for the analyses, will be blinded for allocation group. Only the operator and the participant will be aware of the type of treatment based on the computer-generated allocation table that will be kept at the Trial Master File (TMF) of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control procedure (Active Comparator): Ultrasonic scaling and polishing will be performed every 6 months for subgingival cleaning
  Interventions: Device: Ultrasonic scaler
- Test procedure (Experimental): AIR-FLOW PROPHYLAXIS MASTER with erythritol powder (AIR FLOW Powder Plus) will be used every month for 2 years for subgingival cleaning
  Interventions: Device: Air-Flow Prophylaxis Master

INTERVENTIONS:
Device: Ultrasonic scaler — Ultrasonic scaling for subgingival cleaning every 6 months for 2 years according to the manufacturer's procedures.
  Arms: Control procedure
Device: Air-Flow Prophylaxis Master — AIR-FLOW PROPHYLAXIS MASTER with erythritol powder (AIR FLOW Powder Plus) will be used every month for 2 years for subgingival cleaning according to the manufacturer's procedures.
  Arms: Test procedure

SUMMARY:
Patients with multi-bracketed fixed orthodontic treatment are at increased risk of developing white spot lesions (WSL) and gingivitis. Various preventive strategies have been examined to prevent the development of WSLs. During initial non-surgical periodontal therapy, the use of subgingival air-polishing with erythritol powder has shown promising results in reducing deep pockets and gingival inflammation. The efficacy of its use as monotherapy in preventing WSLs and gingival inflammation in patients during orthodontic treatment, has not yet been tested.

The primary objective of the present study is to compare the effectiveness of an air-polishing device used as monotherapy versus ultrasonic instrumentation (the current gold standard procedure) in preventing white spot lesions (WSL) and gingivitis among young patients undergoing multi-bracketed fixed orthodontic treatment.

DETAILED DESCRIPTION:
This is a randomized clinical study for evaluating the performance of an air-polishing device in preventing WSLs and gingivitis among patients undergoing multi-bracketed fixed orthodontic treatment. The null hypothesis tested is that there is no difference between the air-polishing device and the conventional ultrasonic device in preventing WSLs and gingivitis during orthodontic treatment.

Clinical examination and clinical samples will be taken before, during and after orthodontic treatment. It is a single center study of 3 years duration involving samples of 60 patients attending the Division of Orthodontics for treatment. Half of the participants will be randomly assigned for treatment with the air-polishing device in every orthodontic appointment, meaning once per month, the other half will be treated with a standard ultrasonic scaler every six months. The study duration for each participant will be approximately 2 years. The investigators will then analyze the prevalence of WSLs using the Quantitative light-induced fluorescence (QLF) method. Gingivitis will be evaluated throughout the study by using standard clinical parameters; the antimicrobial efficacy against several known periodontal pathogens and the host-response (inflammatory markers in GCF) will be measured by the qPCR assay and the multiplex immunoassay, respectively. Clinical evaluation and collection of samples for microbial and host response analysis will be performed every 6 months. Incidence of bracket debonding we will be calculated and compared.

ELIGIBILITY:
Inclusion Criteria:

* Subjects about to undergo fixed orthodontic treatment will be invited to participate.
* Age between 12 and 16 years only participants
* Informed written consent obtained by the parents

Exclusion Criteria:

* Clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.),
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the investigation, e.g. due to language problems, psychological disorders, dementia, etc. of the subject
* Participation in another investigation with an investigational drug or another MD within the 30 days preceding and during the present investigation
* Previous enrolment into the current investigation
* Enrolment of the PI, his/her family members, employees and other dependent persons
* History of fixed orthodontic treatment
* Defects on enamel on labial surfaces of the teeth
* Untreated cavitated lesions
* Plaque levels >25%
* Periodontitis
* Multiple missing teeth
* Cleft lip and/or palate or other craniofacial anomalies or syndromes
* Patients taking any regular medication
* Patients with asthmatic problems

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2025-09-11 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Appearance of white spot lesions (WSL) during orthodontic movement with fixed appliances. | 2 years
  Number of participants with white spot lesions appearence during the 2-years period of orthodontic treatment
Appearance on inflammatory lesions during orthodontic treatmnet | 2 years
  Number of participants showing signs of inflammation based on clinical parameters during the 2-year period of orthodontic treatment.
Changes from baseline in clinical parameters | 2 years
  plaque accumulation gingival inflammation pocket probing depth bleeding on probing gingival recessions

SECONDARY OUTCOMES:
Patient acceptance | 2 years
  Visual Analogue Scale (VAS) with 0: very satisfied and 10: unsatisfied
Tooth sensitivity | 2 years
  Visual Analogue Scale (VAS) with 0: no sensitivity and 10: worst senstitivity
Total bacterial counts and counts of 6 periodontal pathogens in subgingival samples from treated pockets | 2 years
  Changes from baseline of microorganisms will be identified and enumerated by laboratory Real-time Polymerase Chain Reaction
Inflammatory markers in GCF from baseline | 2 years
  Changes of the Inflammatory markers in the gingival crevicular fluid (GCF) throughout the study will be analyzed by the Bioplex 200 Suspension array system. The concentration of these markers will be expreseed as pg/ml
Toral tretament time | 2 years
  Treatment time will be recorded at each visit

CONTACTS AND LOCATIONS:
Locations (1):
- University of Geneva, University Clinics of Dental Medicine, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No